CLINICAL TRIAL: NCT04149197
Title: The Down Syndrome Clinical Trials Network (DS-CTN) Study of Alzheimer's Disease in Down Syndrome
Brief Title: Down Syndrome Clinical Trials - Study of Alzheimer's Disease in Down Syndrome
Acronym: LIFE-DSR
Status: Terminated | Type: Observational
Why Stopped: COVID delayed study timelines. Competing studies began enrolling at our sites.
Sponsor: LuMind IDSC Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ADC-059-LIFE-DSR
Record Dates: First submitted 2019-09-26; First posted 2019-11-04 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease in Down Syndrome
Keywords: Down Syndrome; Alzheimer's Disease
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be collected at the baseline, Month 16 and Month 32 visits for banking of plasma for future biomarker studies, which may include analysis of AD biomarkers such as amyloid beta (Aβ) or tau. In addition to biomarker analysis, future genotyping studies may also be conducted. Apolipoprotein E (APOE) (e4 +/-) genotype and other genetic variations are associated with the risk of onset of AD. Therefore, this blood sample collected at baseline, Month 16 and Month 32 will also include banking of buffy coat for future gene analyses which may include APOE testing of e2, e3, and e4 alleles as well as other genes associated with AD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to characterize trajectories of change on the primary outcome measures in this study population through longitudinal collection of measures of cognition, function, behavior, and health status.

DETAILED DESCRIPTION:
The DS-CTN will engage in rigorous, high quality research to better understand AD-DS and the medical needs of this population. The LIFE-DSR study will utilize the DS-CTN network to achieve these goals through evidence-based research and a combination of proven and novel methodologies. The network will initially recruit and employ experts and clinical trial sites who have access to adults with DS and whose focus is on AD-DS.

This trial also aims to develop sensitive and well-validated assessment instruments of cognition, behavior and function appropriate for future clinical trials directed at AD-DS in adults with DS ages 25 and older.

In addition, this LIFE-DSR study will serve as a parent protocol that includes one or more sub-studies, each of which has its own protocol and consent form. These sub-studies will recruit from eligible participants enrolled in this LIFE-DSR protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 years or older
2. Diagnosis of DS, typically supported by karyotype analysis documenting full trisomy for chromosome 21 or complete unbalanced translocation of chromosome 21. Karyotype analysis is not required for study entry
3. Participants, or Legal Authorized Representative, and their study partner if applicable, in the opinion of the investigator, are able to understand and willing to sign written informed consent.
4. Participants must have a study partner who has frequent interaction with the participant on a regular basis, will agree to participate in annual clinic visits, can provide accurate responses to questions about the participant, and facilitate participation in the study visits, in the opinion of site PI or study coordinator.
5. Participant and study partner must be capable of reliably completing study assessments.

Exclusion Criteria Participants and study partners who, in the opinion of the site PI, are not able to complete trial procedures or adhere to the schedule of study assessments will be excluded from study participation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, aged 25 and older, with a diagnosis of DS, typically supported by karyotype analysis documenting full trisomy for chromosome 21 or complete unbalanced translocation of chromosome 21.
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Cognitive Measure | through study completion, an average of 2 years
  Severe Impairment Battery (SIB) with Shoebox Test. If the participant achieves a score 60 or above on the SIB, the Down Syndrome Mental Status Examination (DS-MSE) will also be administered. Subscale Ranges:
  Social Interaction - 0 - 6 Orientation - 0 - 8 Visuospatial Ability - 0 - 8 Construction - 0 - 12 Language - 0 - 56 Memory - 0 - 16 Praxis - 0 - 8 Attention - 0 - 15 Orienting to name - 0 - 4
  Higher scores reflect better performance for each subscale. Scores above 60 mean the participant completes the Shoebox Memory Test.
Functional Measure | through study completion, an average of 2 years
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Vineland-3 is an adaptive behavior measure used to assess intellectual/developmental/other disabilities. Total score range: 0 - 140
  Expressive Communication: 0 - 98 49 questions - range: 0 - 2 per Q Written Communication: 0 - 76 38 questions - range: 0 - 2 per Q Personal Daily Living Skills - 0 - 110 55 questions - range: 0 - 2 per Q
Behavioral Measure | through study completion, an average of 2 years
  Dementia Questionnaire for People with Learning Disabilities (DLD) - Measures specific cognitive and functional deterioration as a result of dementia, and functional deterioration as a result of severe sensory or psychiatric problems. Range of total possible scores: 0 - 100 50 Questions with a possible range of 0 - 2 per question. Higher scores reflect worse performance.
  Score Calculation:
  Categories are mixed throughout the questionnaire. To calculate the score at the end, scores on each page are added up and categorizes into Cognitive Scores, or SCS (categories 1 - 3: Short-term memory, Long-term memory, and Spatial & Temporal Orientation) and Social Scores, or SOS (Categories 4 - 8: Speech, Practical Skills, Mood, Activity & Interest, Behavioral Disturbance).
Health Measures | through study completion, an average of 2 years
  New-onset seizures or significantly increased frequency of seizures
Behavioral Measure | through study completion, an average of 2 years
  Neuropsychiatric Inventory (NPI) - Neuropsychiatric Inventory (NPI) evaluates both the frequency and severity of 10 neuropsychiatric features, including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability and lability, and aberrant motor behavior, as well as evaluates sleep and appetite/eating disorders. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously). Severity assessments range from 1 (mild) to 3 (severe). The score for each subscale is the product of severity and frequency and the total score is the sum of all subscales.

SECONDARY OUTCOMES:
Exploratory Outcome Measure Preliminary composite measure from the scales being used in LIFE-DSR | through study completion, an average of 2 years
  To derive a preliminary composite measure from the scales being used in LIFE-DSR that is most sensitive to change in this population and which can be validated in a future prospective study. If the participant achieves a score 60 or above on the SIB, the Down Syndrome Mental Status Examination (DS-MSE) will also be administered. The maximum score is 100.
Exploratory Outcome Measure Novel multi-domain instrument for AD-DS development | through study completion, an average of 2 years
  To integrate and further validate a novel and highly sensitive multidomain instrument for AD-DS upon its completion (Professor A. Strydom, Kings College, London). This instrument is being developed under a separate protocol and upon its validation will be integrated into LIFE-DSR to evaluate its responsiveness to change in clinically important domains.
Exploratory Outcome Measure Potential Screening Measures | through study completion, an average of 2 years
  Individual subscales from the larger test batteries included in the LIFE-DSR Primary Outcome Measures, Severe Impairment Battery (SIB) with Shoebox Test, the Down Syndrome Mental Status Examination (DS-MSE), NPI, and Vineland3. These could then be further validated in a future prospective study.
  SIB - Social Interaction - 0 - 6 Orientation - 0 - 8 Visuospatial Ability - 0 - 8 Construction - 0 - 12 Language - 0 - 56 Memory - 0 - 16 Praxis - 0 - 8 Attention - 0 - 15 Orienting to name - 0 - 4
  Scores above 60 mean the participant completes the Shoebox Memory Test.
  Vineland-3 -Total score range: 0 - 140
  DLD - Questions with a possible range of 0 - 2 per question. Higher scores reflect worse performance.
  NPI - The score for each subscale is the product of severity and frequency and the total score is the sum of all subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Lois Kelly, Study Director — LuMind IDSC Foundation
Locations (14):
- United States (14):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University California Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Health, Park Ridge, Illinois
  - Kansas University Medical Center, Fairway, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No